CLINICAL TRIAL: NCT03609580
Title: Post-operative Urinary Retention (POUR) Following Thoracic Surgery
Acronym: POUR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO#2017-0687
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urinary Retention
Keywords: post operative urinary retention; inability to urinate; urinary retentions; lung cancer; VATs; Robotic Lung Surgery; lung resections
MeSH Terms: conditions — Urinary Retention; Lung Neoplasms | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 week Pre-operative Tamsulosin administration (Experimental)
  Interventions: Drug: Tamsulosin - 1 week
- 3 days Pre-operative Tamsulosin administration (Experimental)
  Interventions: Drug: Tamsulosin - 3 days

INTERVENTIONS:
Drug: Tamsulosin - 1 week — The investigators hypothesize that pre-operative administration of Tamusolin (Flomax, 0.4mg/day x 1 week), with ongoing use post-operatively until normal voiding resumes, will result in a significant decrease in the incidence of POUR after a thoracic surgical procedure.
  Arms: 1 week Pre-operative Tamsulosin administration
Drug: Tamsulosin - 3 days — The investigators hypothesize that pre-operative administration of Tamusolin (Flomax, 0.4mg/day x 3 days), with ongoing use post-operatively until normal voiding resumes, will result in a significant decrease in the incidence of POUR after a thoracic surgical procedure.
  Arms: 3 days Pre-operative Tamsulosin administration

SUMMARY:
Inability to urinate a common complication that happens to many patients after a surgery, especially in men over 60 years of age who undergo surgery on their chest. Urinary retention is uncomfortable, increases anxiety, increases hospital length of stay, and leads to more procedures such as putting in a bladder catheter (Foley). This is uncomfortable, and can lead to bleeding, infection, damage to the urethra and/or bladder and bladder spasm. The goal of this study is to attempt to prevent inability to urinate by giving patients a medication called Flomax (Tamusolin) every day beginning a week before surgery. That medication relaxes the prostate. It's approved by the Food and Drug Administration (FDA) to improve urinary flow in those with enlarged prostates. It is also commonly used in patients with bladder problems due to inability to urinate who have required a Foley.

DETAILED DESCRIPTION:
Post-operative urinary retention (POUR) in older men who undergo a thoracic surgical procedure occurs in a significant proportion of patients (25% at Hackensack University Medical Center in men >60) and is a significant management problem. Typically, this complication needs to be treated with placement of a bladder catheter (foley). In addition to the discomfort of placing a foley in an awake patient, these patients are at a significantly increased risk of a catheter associated urinary tract infection (CAUTI), potential genito-urinary injury during the placement, and bladder muscle damage due to distention.

The goal of this study is to investigate whether the use of Tamusolin could lower the high incidence of POUR in older men undergoing a thoracic surgical procedure.

The investigators hypothesize that pre-operative administration of Tamusolin (Flomax, 0.4mg/day x 1 week), with ongoing use post-operatively until normal voiding resumes, will result in a significant decrease in the incidence of POUR after a thoracic surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

Males

≥50 years old Planned surgical procedure of a minimally invasive thoracic surgical procedure (wedge resection, segmentectomy, lobectomy, pleural biopsy, or pleurodesis) Surgery scheduled more than 3 days from the time of consent

Exclusion Criteria:

* Using Flomax already
* Allergy to Flomax or sulfa drugs
* Current use of alpha blockers or alpha agonists
* Resting systolic blood pressure <100
* Orthostatic hypotension of >20mm Hg (millimeters of mercury) Systolic and/or 10mm Hg diastolic pressure from sitting to standing (after 2 minutes of standing) as measured at the time of consent
* Known diagnosis of congestive heart failure and valvular heart disease
* History of prostate surgery (prostatectomy, trans-urethral resection)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 127 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Volume of urine (cc) post thoracic surgery in patients that received Flomax, 0.4mg/day for a week before surgery | 8 hours
  The absence of voiding naturally after undergoing thoracic surgery needing an intervention as a Foley catheter or a catheterization. Documentation for first void, Post bladder scan showing more that 300cc of residual urine in the bladder (failure to urinate), or following spontaneous urination if there is more than 300cc of residual urine in the bladder (inadequate urination)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mansour, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Daniel Mansour, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No